CLINICAL TRIAL: NCT05959161
Title: Study on Brain Network Mechanism of Deep Brain Stimulation for Parkinson's （A Retrospective Study）
Brief Title: Study on Brain Network Mechanism of Deep Brain Stimulation for Parkinson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Guangrui Zhao, Associate Professor of Neurosurgery, Huanhu Hospital, Tianjin University, Tianjin Huanhu Hospital
Other Study IDs: TianjinHH
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease; Deep Brain Stimulation; Non-motor Symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- improvement and no improvement: We observed whether the symptoms of patients improved after DBS surgery and divided them into groups.
  Interventions: Procedure: DBS
- imp+ and imp-
  Interventions: Procedure: DBS

INTERVENTIONS:
Procedure: DBS — We observed the prognostic changes of patients after DBS surgery

SUMMARY:
As a surgical intervention, DBS can effectively relieve PD tremor, rigidity, bradykinesia and other symptoms. How to better screen patients suitable for DBS treatment and conduct reasonable preoperative and postoperative evaluation is crucial to judge the treatment effect and prognosis. The clinical symptom evaluation of PD patients can be divided into motor symptom evaluation and non-motor symptom evaluation. The motor symptoms of PD patients were evaluated by UPDRS III. The evaluation of non-motor symptoms in PD patients was mainly divided into three aspects: cognitive status, emotional status, and sleep status. Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA) were used to assess the cognitive status of PD patients. The Hamilton Depression Scale (HAMD) was used to assess the patients' depression status. The Hamilton Anxiety Scale (HAMA) was used to assess the patients' anxiety status. The PD Sleep Scale 2nd version, The PD Sleep Scale 2nd version, PDSS - 2), and rem Sleep Behavior Disorder Questionnaire (sweet HK) (Rapid Eye Movement Sleep behaviors Disorder Questionnaire - Hong Kong, RBDQ - HK) to assess Sleep conditions.

ELIGIBILITY:
Inclusion Criteria:The clinical diagnosis of PD is consistent with the United Kingdom Parkinson's Disease Society Brain Bank criteria, with disease duration over 5 years, age under 75, acute levodopa motor response ≥30%, and indication for STN-DBS. -

Exclusion Criteria: patients with severe cognitive impairment, severe psychiatric disorders, acute levodopa motor response less than 30%, atypical parkinsonism, and contraindications to surgery -

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary Parkinson's disease were followed up for 1 year after deep brain stimulation, and the imaging data were intact
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
motor symptom | 2023.1 to 2025.12
  UPDRS III score changes

IPD SHARING:
Plan to Share IPD: Undecided